CLINICAL TRIAL: NCT01147978
Title: Impact of a Proactive Strategy of Communication With Patients Hospitalized in ICU and Their Families With the Aim of Reducing Their Anxious and Depressive Symptoms and Their Post Traumatic Stress Symptoms
Brief Title: Proactive Communication Strategy in Intensive Care Unit and Post Traumatic Stress Symptoms
Acronym: FAMIREAXV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: University Paris 7 - Denis Diderot (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K070101; ID RCB / 2007-A01044-49 (Other Grant/Funding Number: APHP)
Record Dates: First submitted 2010-06-18; First posted 2010-06-22 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Critically Ill Patients
Keywords: ICU; Anxiety; Depression; PTSD
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- End of ICU stay conference (Experimental): Conference with patient and proxies, senior physician and nurse regarding the ICU stay and the orientation of the patient
  Interventions: Behavioral: End of ICU stay conference
- Usual Procedure (No Intervention): Usual discharge procedure from the ICU

INTERVENTIONS:
Behavioral: End of ICU stay conference — Conference with patient and proxies, senior physician and nurse regarding the ICU stay and the orientation of the patient
  Arms: End of ICU stay conference

SUMMARY:
The investigators propose an interventional multicentric (23 ICUs) study measuring the impact of a consultation at the end of ICU stay for the patients and his/her families on the prevalence of symptoms of PTSD and anxiety or depression 3 months and one year after discharge. Patients will be randomly assigned to a intervention or control group. In the intervention group, the patient and his/her family will benefit from an conference by the intensivist at the end of the ICU stay, regarding information about the progress of his stay in ICU, his orientation after discharge, the possibility of consulting a GP, etc. Patients and proxies will be interviewed by phone three months and one year after discharge from ICU. Main instruments are Hospital Anxiety and Depression Scale, and Impact of Events Scale Revised.

DETAILED DESCRIPTION:
There are many risk factors of stress for a patient during a stay in Intensive care unit. This stress can be responsible for psychiatric symptoms hindering seriously the quality of life of the patient in the months following discharge from ICU. Survivors of ICU suffer from traumatic memories (nightmares, acute anxiety), who can be associated to post traumatic stress disorder (PTSD) or of anxious and depressive symptoms. Prevalence of PTSD in the months following ICU stay is estimated between 14 and 41 %, that of the symptoms of anxiety between 12 % and 47 %, and that of the symptoms of depression between 10 % and 30 %. Recent studies showed that these symptoms could concern several thousand patients every year in France.

We propose an interventional multicentric (23 ICUs) study measuring the impact of a consultation at the end of ICU stay for the patients and his/her families on the prevalence of symptoms of PTSD and anxiety or depression 3 months and one year after discharge.

Patients will be randomly assigned to a intervention or control group. In the intervention group, the patient and his/her family will benefit from an conference by the intensivist at the end of the ICU stay, regarding information about the progress of his stay in ICU, his orientation after discharge, the possibility of consulting a general practitioner (GP), etc. The family, if present, will be invited to attend the conference. In the control group, patients will be cared in a usual way (without end of stay conference) as it is made in all the intensive care units in France. Inclusion criteria are 1) patient alive at the end of ICU stay, 2) Age > 18 years, 3) more than 48 hours of mechanical ventilation 4) accepting to be called back 3-month and on one year after discharge of ICU. Exclusion criteria are 1) Chronic cognitive deterioration before ICU admission, 2) inclusion in another interventional randomized essay 3) non French-speaking patients, 4) impossibility to agree 5) End of life situation (survival at 3 months very improbable), 6) deaf-dumb patients. Patients and proxies will be interviewed by phone three months and one year after discharge from ICU. Main instruments are Hospital Anxiety and Depression Scale, and Impact of Events Scale Revised. Number of patients to include takes into account an estimated prevalence of PTSD of 20 %, and the impact expected from the intervention is to obtain 10 % of PTSD in the intervention group. With a beta power of 90 % and a risk of 5 %, number of patients needed three months after discharge is 438 (219 in every group), i.e 525 patients (263 in every arm because of the late deaths and lost sight). This study should supply updated and relevant data on prevalence and risk factors of symptoms of PTSD and Anxiety-depression three months and one year after discharge from ICU. Furthermore, we propose an intervention that could demonstrate that a brief and easily reproducible communication strategy could significantly reduce prevalence of PTSD and anxiety-depression for patients and their families after discharge from ICU

ELIGIBILITY:
Inclusion Criteria:

* patient alive at the end of ICU stay
* age > 18 years
* more than 48 hours of mechanical ventilation
* accepting to be called back 3-month and on one year after discharge of ICU.

Exclusion Criteria:

* chronic cognitive deterioration before ICU admission
* inclusion in another interventional randomized essay
* non French-speaking patients
* impossibility to agree for participation
* end of life situation (survival at 3 months very improbable)
* deaf-dumb patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2009-04; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Symptoms of PTSD in ICU patients | three months after discharge from ICU

SECONDARY OUTCOMES:
Symptoms of PTSD, anxiety, and depression in ICU patients | three months after discharge from ICU
Symptoms of PTSD, anxiety, and depression in ICU patients | one year after discharge from ICU
Symptoms of PTSD, anxiety, and depression in families | three months after discharge from ICU
Symptoms of PTSD, anxiety, and depression in families | one year after discharge from ICU

CONTACTS AND LOCATIONS:
Overall Officials: Elie AZOULAY, MD PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Medical ICU, Paris, Paris, France